CLINICAL TRIAL: NCT03629886
Title: Safety and Protective Effect Study of GSK Biologicals' Human Papillomavirus (Types 16, 18) Vaccine, Adsorbed (GSK580299) in Healthy Female Subjects From the HPV-039 Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205779
Record Dates: First submitted 2018-07-24; First posted 2018-08-14 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Adults; Human Papillomavirus (HPV); Cervical cancer; Safety
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacc-039 Group (No Intervention): Healthy Chinese female subjects, above 26 years of age at study entry, who previously received HPV vaccine in HPV-039 study (NCT00779766), underwent cervical sample collection and didn't receive any vaccine in the current study.
- Vacc-092 Group (Experimental): Healthy Chinese female subjects, above 26 years of age at study entry, who previously received placebo (control group) in HPV-039 study (NCT00779766), were intended to receive HPV vaccine in the current study and were to provide cervical samples before HPV vaccination.
  Interventions: Biological: HPV (Types 16, 18) Vaccine, Adsorbed

INTERVENTIONS:
Biological: HPV (Types 16, 18) Vaccine, Adsorbed — Three doses of Human Papillomavirus (Types 16, 18) Vaccine, Adsorbed administered intramuscularly in the deltoid region of the upper arm, according to a 0, 1, 6-month schedule.
  Arms: Vacc-092 Group

SUMMARY:
This study was designed to enable all subjects who received placebo in the HPV-039 study (NCT00779766), to also receive GSK Biologicals' Human Papillomavirus (Types 16, 18) Vaccine, Adsorbed. Safety data in terms of serious adverse events (SAEs), any adverse events (AEs)/SAEs leading to premature discontinuation of the study, potential immune mediated diseases (pIMDs) and pregnancies (and their outcomes) were collected during the study period.

In addition, this study assessed the long term protective effect of the vaccine, in an exploratory manner, in terms of rates of HPV-related (vaccine type) incident cervical infection up to approximately 10 years after vaccination in subjects who participated in HPV-039 study (NCT00779766).

DETAILED DESCRIPTION:
Treatment allocation depended on the randomization in the previous study i.e. only the subjects from the control group of HPV-039 study received HPV vaccination in the current study. Subjects who previously received the Human Papillomavirus (Types 16, 18) Vaccine, Adsorbed in HPV-039 study did not receive vaccination in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* Subjects previously enrolled in the HPV-039 study.
* Subjects with negative pregnancy test at Visit 1.

Additional inclusion criteria for subjects of HPV group undergoing vaccination ONLY:

* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Previous vaccination against HPV outside of study HPV-039.

Additional exclusion criteria for subjects of HPV group undergoing vaccination ONLY:

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine/product not foreseen by the study protocol in the period starting 30 days before and after each dose of vaccine administration, with the exception of administration of routine vaccines e.g. meningococcal, hepatitis B, hepatitis A, inactivated influenza up to eight days before and after each dose of study vaccine. Enrolment will be deferred until the subject is outside of the specified window.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Previous administration of MPL or AS04 adjuvant.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Cancer or autoimmune disease under treatment.
* Hypersensitivity to latex.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.0°C. The preferred location for measuring temperature in this study will be the axilla.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Pregnant or breastfeeding. Subjects must be at least three months post-pregnancy and not breastfeeding to enter the study.
* Females planning to become pregnant or planning to discontinue contraceptive precautions during the vaccination phase of the study, i.e. up to two months after the last vaccine dose.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6051 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- China (4):
  - GSK Investigational Site, Jintan, Jiangsu
  - GSK Investigational Site, Lianshui, Jiangsu
  - GSK Investigational Site, Xuzhou, Jiangsu
  - GSK Investigational Site, Yancheng, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Zhao F, Jastorff A, Hong Y, Hu S, Chen W, Xu X, Zhu Y, Zhu J, Zhang X, Zhang W, Xu D, Wang D, Tang R, Sun Y, Shen Y, Pan Q, Yin J, Liu D, Liu B, Karkada N, Jiang C, Cui J, Chen F, Bi J, Bao Y, Zhou X, Cartier C, Hu Y, Borys D. Safety of AS04-HPV-16/18 vaccine in Chinese women aged 26 years and older and long-term protective effect in women vaccinated at age 18-25 years: A 10-year follow-up study. Asia Pac J Clin Oncol. 2023 Aug;19(4):458-467. doi: 10.1111/ajco.13833. Epub 2022 Sep 13. PMID 36101936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 centers in China.
Period: Overall Study
Arm/Group | Vacc-039 Group | Vacc-092 Group
Started | 1671 | 1866
Completed | 1671 | 1686
Not Completed | 0 | 180
Not completed — Migrated / moved from the study area | 0 | 55
Not completed — Consent withdrawal, not due to an AE | 0 | 50
Not completed — Study vaccine not administrated | 0 | 3
Not completed — Didn't meet inclusion/exclusion criteria | 0 | 28
Not completed — Refused vaccination step of the study | 0 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vacc-039 Group | Vacc-092 Group | Total
Number analyzed (Participants) | 1671 | 1866 | 3537
Age, Customized [Count of Participants; unit: Participants]
  Between 24 and 64 years | 1671 | 1866 | 3537
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1671 | 1866 | 3537
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Chinese Heritage | 1671 | 1866 | 3537

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to Study Vaccine in Vacc-092 Group
Description: SAEs assessed include any untoward medical occurrence that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Related SAEs are those SAEs assessed by the investigator as related to vaccination in the study.
Time Frame: During the entire study period (Day 1-Month 12)
Population: Analysis was performed on all subjects who received at least one dose of HPV vaccine (Vacc-092 Group) in the current study and for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Vacc-092 Group
Number analyzed (Participants) | 1791
Participants | 0

2. Secondary Outcome: Number of Subjects With Potential Immune Mediated Diseases (pIMDs) in Vacc-092 Group
Description: pIMDS are a subset of adverse events (AEs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which might or might not have an autoimmune aetiology.
Time Frame: During the entire study period (Day 1-Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vacc-092 Group
Number analyzed (Participants) | 1791
Participants | 1

3. Secondary Outcome: Number of Pregnant Subjects Reported With Outcomes of Pregnancy in Vacc-092 Group
Description: Pregnancy is the term used to describe the period in which a fetus develops inside a woman's womb or uterus. The subjects with confirmed pregnancies were followed up to determine the outcomes of the reported pregnancies. Outcomes of the reported pregnancies were: Live infant no apparent Congenital Anomaly (CA), Live infant CA, Elective termination no apparent CA, Elective termination CA, Spontaneous abortion no apparent CA, Spontaneous abortion CA, Stillbirth no apparent CA, Stillbirth CA, Ectopic pregnancy, Molar pregnancy, Lost to follow-up & Pregnancy ongoing.
Time Frame: During the entire study period (Day 1-Month 12)
Population: Analysis was performed on pregnant subjects from the Vacc-092 Group in the current study and for whom pregnancy outcomes data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Vacc-092 Group
Number analyzed (Participants) | 10
Participants
  Live infant no apparent CA | 2
  Live infant CA | 0
  Elective termination no apparent CA | 8
  Elective termination CA | 0
  Spontaneous abortion no apparent CA | 0
  Spontaneous abortion CA | 0
  Stillbirth no apparent CA | 0
  Stillbirth CA | 0
  Ectopic pregnancy | 0
  Molar pregnancy | 0
  Lost to follow-up | 0
  Pregnancy ongoing | 0

4. Secondary Outcome: Number of Subjects With SAEs in Vacc-092 Group
Description: SAEs assessed include any untoward medical occurrence that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (Day 1-Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vacc-092 Group
Number analyzed (Participants) | 1791
Participants | 1

5. Secondary Outcome: Number of Subjects With Any Adverse Events or Serious Adverse Events (AE/SAE) Leading to Premature Discontinuation From the Study in Vacc-092 Group
Description: AEs assessed include any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. SAEs assessed include any untoward medical occurrence that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any is defined as the occurrence of any unsolicited AE/SAE regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (Day 1-Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vacc-092 Group
Number analyzed (Participants) | 1791
Participants | 0

6. Secondary Outcome: Number of Subjects With SAEs Related to Study Participation in All Study Groups
Description: SAEs assessed include any untoward medical occurrence that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Related SAEs are those SAEs assessed by the investigator as activities related to study participation and not by study vaccine (e.g. SAEs due to invasive tests).
Time Frame: During the entire study period (Day 1-Month 12)
Population: Analysis was performed on the Total Enrolled Set, which included all subjects enrolled in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vacc-039 Group | Vacc-092 Group
Number analyzed (Participants) | 1671 | 1866
Participants | 0 | 0

7. Secondary Outcome: Incidence Rates of Incident Cervical Infection With HPV-16 and/or HPV-18 (by PCR) in HPV DNA Negative and Seronegative Subjects at Baseline in All Study Groups
Description: The incidence rate (n/T) of incident cervical infection with HPV-16 and/or HPV-18 (per 100 Person-years rate) was calculated as the number of subjects reporting at least one event (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Cervical infection caused by HPV Types 16 and 18 was assessed by detecting HPV DNA using Polymerase Chain Reaction (PCR). For single HPV type: Subjects DNA negative at Month 0 and seronegative at Month 0 for the corresponding HPV type in study HPV 039 (NCT00779766). For combined HPV types: Subjects DNA negative at Month 0 and seronegative at Month 0 for at least one HPV type (subjects were in the analysis of at least one single type) in study HPV 039 (NCT00779766).
Time Frame: From Month 0 in HPV-039 (NCT00779766) study [at the Day after Dose 1 (out of 3 doses administered in HPV-039)] until Month 120 (corresponding to Day 1 in the current study)
Population: Analysis was performed on all subjects who participated in the current study, who were HPV DNA negative and seronegative at baseline [at Month 0 in HPV-039 (NCT00779766) study] and who had cervical samples collected data.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Vacc-039 Group | Vacc-092 Group
Number analyzed (Participants) | 1486 | 1678
events per 100 person-years
  HPV-16: number analyzed (Participants) | 1154 | 1273
  HPV-16 | 0.13 [0.07 to 0.21] | 0.8 [0.65 to 0.98]
  HPV-18: number analyzed (Participants) | 1383 | 1554
  HPV-18 | 0.07 [0.03 to 0.13] | 0.43 [0.33 to 0.55]
  HPV-16/18 | 0.16 [0.10 to 0.24] | 0.94 [0.79 to 1.11]
Statistical Analysis 1: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-16 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=1963). Those subjects were or were not enrolled in the current study, were HPV DNA negative and seronegative subjects at baseline and had cervical samples collected data; Test type: Other — The IR (n/T) of incident cervical infection with HPV-16 (per 100 Person-years rate) was calculated as the number of subjects reporting at least one event (n), over the sum of follow-up period expressed in years (T), and multiplied by 100 and 95% Confidence Intervals (CI) were used for calculation; Incidence rate per 100 Person-years = 0.15, 95% CI 2-sided [0.09 to 0.23]
Statistical Analysis 2: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-16 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=1917). Those subjects were or were not enrolled in the current study, were HPV DNA negative and seronegative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 7, analysis 1]; Incidence rate per 100-Person years = 0.88, 95% CI 2-sided [0.73 to 1.05]
Statistical Analysis 3: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-18 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2356). Those subjects were or were not enrolled in the current study, were HPV DNA negative and seronegative subjects at baseline and had cervical samples collected data; Test type: Other — The IR (n/T) of incident cervical infection with HPV-18 (per 100 Person-years rate) was calculated as the number of subjects reporting at least one event (n), over the sum of follow-up period expressed in years (T), and multiplied by 100 and 95% Confidence Intervals (CI) were used for calculation; Incidence rate per 100-Person years = 0.09, 95% CI 2-sided [0.05 to 0.15]
Statistical Analysis 4: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-18 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2357). Those subjects were or were not enrolled in the current study, were HPV DNA negative and seronegative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 7, analysis 3]; Incidence rate per 100-Person years = 0.44, 95% CI 2-sided [0.35 to 0.56]
Statistical Analysis 5: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-16/18 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2534). Those subjects were or were not enrolled in the current study, were HPV DNA negative and seronegative subjects at baseline and had cervical samples collected data; Test type: Other — The IR (n/T) of incident cervical infection with HPV-16 and/or HPV-18 (per 100 Person-years rate) was calculated as the number of subjects reporting at least one event (n), over the sum of follow-up period expressed in years (T), and multiplied by 100 and 95% Confidence Intervals (CI) were used for calculation; Incidence rate per 100 Person-years = 0.20, 95% CI 2-sided [0.14 to 0.27]
Statistical Analysis 6: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-16/18 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2547). Those subjects were or were not enrolled in the current study, were HPV DNA negative and seronegative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 7, analysis 5]; Incidence rate per 100 Person-years = 1.02, 95% CI 2-sided [0.88 to 1.18]

8. Secondary Outcome: Incidence Rates of Incident Cervical Infection With HPV-16 and/or HPV-18 (by PCR) in HPV DNA Negative Subjects at Baseline, Regardless of Initial Serostatus in All Study Groups
Description: The incidence rate (n/T) of incident cervical infection with HPV-16 and/or HPV-18 (per 100 Person-years rate) was calculated as the number of subjects reporting at least one event (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Cervical infection caused by HPV Types 16 and 18 was assessed by detecting HPV DNA using Polymerase Chain Reaction (PCR). For single HPV type: Subjects DNA negative at Month 0 for the corresponding HPV type in study HPV-039 (NCT00779766). For combined HPV types: Subjects DNA negative at Month 0 for at least one HPV type (subjects were in the analysis of at least one single type) in study HPV-039 (NCT00779766).
Time Frame: as for outcome 7
Population: Analysis was performed on all subjects who participated in the current study, who were HPV DNA negative at baseline [at Month 0 in HPV-039 (NCT00779766) study] regardless of initial serostatus and who had cervical samples collected data.
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Vacc-039 Group | Vacc-092 Group
Number analyzed (Participants) | 1647 | 1841
events per 100 person-years | 0.22 [0.15 to 0.3] | 1.1 [0.95 to 1.27]
Statistical Analysis 1: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-16/18 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2818). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 7, analysis 5]; Incidence rate per 100-Person years = 0.25, 95% CI 2-sided [0.19 to 0.33]
Statistical Analysis 2: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of HPV-16/18 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2815). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 7, analysis 5]; Incidence rate per 100-Person years = 1.21, 95% CI 2-sided [1.06 to 1.37]

9. Secondary Outcome: Incidence Rates of Incident Cervical Infection With Any Oncogenic HPV Type or Combination of Oncogenic HPV Types in HPV DNA Negative Subjects at Baseline, Regardless of Initial Serostatus in All Study Groups
Description: The IR (n/T) of incident cervical infection with any oncogenic HPV type or combination of oncogenic HPV types (per 100 Person-years rate) was calculated as the number of subjects reporting at least one event (n) in a group (assessed by detecting HPV DNA using PCR), over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Oncogenic HPV types assessed were HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68. HRW-HPV = High-risk (oncogenic) HPV types without HPV-16 or HPV-18: HPV-31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68. HR-HPV = High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68. For single type: Subjects DNA negative at Month 0 for the corresponding HPV type in NCT00779766 study. For combined types: Subjects DNA negative at Month 0 for at least one HPV type (subjects were in the analysis of at least 1 single type) in NCT00779766 study.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Vacc-039 Group | Vacc-092 Group
Number analyzed (Participants) | 1650 | 1842
events per 100 person-years
  HPV-16: number analyzed (Participants) | 1597 | 1796
  HPV-16 | 0.14 [0.09 to 0.22] | 0.79 [0.66 to 0.93]
  HPV-18: number analyzed (Participants) | 1629 | 1827
  HPV-18 | 0.08 [0.04 to 0.13] | 0.45 [0.36 to 0.56]
  HPV-31: number analyzed (Participants) | 1632 | 1837
  HPV-31 | 0.25 [0.17 to 0.34] | 0.46 [0.36 to 0.57]
  HPV-33: number analyzed (Participants) | 1633 | 1827
  HPV-33 | 0.29 [0.21 to 0.39] | 0.39 [0.3 to 0.5]
  HPV-35: number analyzed (Participants) | 1642 | 1836
  HPV-35 | 0.20 [0.14 to 0.29] | 0.32 [0.24 to 0.42]
  HPV-39: number analyzed (Participants) | 1620 | 1823
  HPV-39 | 0.71 [0.58 to 0.86] | 0.78 [0.65 to 0.93]
  HPV-45: number analyzed (Participants) | 1638 | 1835
  HPV-45 | 0.13 [0.08 to 0.2] | 0.22 [0.16 to 0.31]
  HPV-51: number analyzed (Participants) | 1628 | 1815
  HPV-51 | 0.94 [0.79 to 1.11] | 0.93 [0.79 to 1.09]
  HPV-52: number analyzed (Participants) | 1600 | 1776
  HPV-52 | 1.67 [1.47 to 1.9] | 1.67 [1.47 to 1.88]
  HPV-56: number analyzed (Participants) | 1636 | 1819
  HPV-56 | 0.49 [0.39 to 0.62] | 0.52 [0.42 to 0.64]
  HPV-58: number analyzed (Participants) | 1633 | 1815
  HPV-58 | 0.44 [0.34 to 0.56] | 0.61 [0.5 to 0.74]
  HPV-59: number analyzed (Participants) | 1648 | 1828
  HPV-59 | 0.29 [0.21 to 0.38] | 0.32 [0.24 to 0.42]
  HPV-66: number analyzed (Participants) | 1636 | 1813
  HPV-66 | 0.57 [0.46 to 0.7] | 0.63 [0.52 to 0.77]
  HPV-68: number analyzed (Participants) | 1633 | 1825
  HPV-68 | 0.48 [0.37 to 0.6] | 0.55 [0.44 to 0.67]
  HPV-31/33/45 | 0.58 [0.47 to 0.71] | 0.93 [0.79 to 1.09]
  HPV-16/18/33/31/45 | 0.8 [0.66 to 0.96] | 1.91 [1.7 to 2.14]
  HRW-HPV | 4.73 [4.35 to 5.13] | 5.13 [4.75 to 5.53]
  HR-HPV | 4.85 [4.47 to 5.26] | 5.56 [5.16 to 5.98]
Statistical Analysis 1: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-16 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2718). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — The IR (n/T) of incident cervical infection with any oncogenic HPV type or combination of oncogenic HPV types (per 100 Person-years rate) was calculated as the number of subjects reporting at least one event (n) in a group (assessed by detecting HPV DNA using PCR), over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100 and 95% Confidence Intervals (CI) were used for calculation; Incidence rate per 100-Person years = 0.17, 95% CI 2-sided [0.11 to 0.24]
Statistical Analysis 2: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-16 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2722). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.85, 95% CI 2-sided [0.72 to 0.99]
Statistical Analysis 3: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-18 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2781). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.10, 95% CI 2-sided [0.06 to 0.15]
Statistical Analysis 4: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-18 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2781). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.47, 95% CI [0.38 to 0.58]
Statistical Analysis 5: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-31 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2786). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.21, 95% CI 2-sided [0.15 to 0.28]
Statistical Analysis 6: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-31 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2782). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.48, 95% CI 2-sided [0.39 to 0.59]
Statistical Analysis 7: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-33 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2779). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.25, 95% CI 2-sided [0.18 to 0.33]
Statistical Analysis 8: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-33 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2784). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.41, 95% CI 2-sided [0.33 to 0.51]
Statistical Analysis 9: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-35 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2806). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.30, 95% CI 2-sided [0.23 to 0.39]
Statistical Analysis 10: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-35 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2803). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.36, 95% CI 2-sided [0.28 to 0.46]
Statistical Analysis 11: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-39 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2759). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.88, 95% CI [0.75 to 1.02]
Statistical Analysis 12: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-39 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2773). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.79, 95% CI 2-sided [0.67 to 0.93]
Statistical Analysis 13: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-45 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2794). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.11, 95% CI 2-sided [0.07 to 0.16]
Statistical Analysis 14: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-45 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N= 2802). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.21, 95% CI 2-sided [0.15 to 0.28]
Statistical Analysis 15: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-51 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2753). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 1.02, 95% CI 2-sided [0.88 to 1.18]
Statistical Analysis 16: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-51 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2756). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 1.18, 95% CI 2-sided [1.03 to 1.34]
Statistical Analysis 17: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-52 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2666). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 1.67, 95% CI 2-sided [1.48 to 1.87]
Statistical Analysis 18: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-52 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2663). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 1.80, 95% CI 2-sided [1.61 to 2.00]
Statistical Analysis 19: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-56 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2783). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.61, 95% CI 2-sided [0.50 to 0.73]
Statistical Analysis 20: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-56 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2779). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.64, 95% CI 2-sided [0.53 to 0.76]
Statistical Analysis 21: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-58 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2772). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.51, 95% CI 2-sided [0.42 to 0.62]
Statistical Analysis 22: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-58 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2768). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.65, 95% CI [0.55 to 0.77]
Statistical Analysis 23: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-59 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2814). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.31, 95% CI 2-sided [0.24 to 0.40]
Statistical Analysis 24: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-59 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2797). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.36, 95% CI 2-sided [0.28 to 0.45]
Statistical Analysis 25: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-66 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2779). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.62, 95% CI 2-sided [0.51 to 0.74]
Statistical Analysis 26: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-66 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2763). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.64, 95% CI 2-sided [0.54 to 0.77]
Statistical Analysis 27: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-68 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2775). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.56, 95% CI [0.46 to 0.68]
Statistical Analysis 28: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-68 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2785). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.59, 95% CI 2-sided [0.49 to 0.71]
Statistical Analysis 29: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-31/33/45 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2823). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.50, 95% CI 2-sided [0.41 to 0.61]
Statistical Analysis 30: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-31/33/45 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2824). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.97, 95% CI 2-sided [0.84 to 1.12]
Statistical Analysis 31: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-16/18/33/31/45 incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2823). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 0.75, 95% CI 2-sided [0.63 to 0.88]
Statistical Analysis 32: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HPV-16/18/33/31/45 incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2825). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 2.11, 95% CI 2-sided [1.91 to 2.33]
Statistical Analysis 33: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HRW-HPV incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2823). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 5.13, 95% CI 2-sided [4.79 to 5.49]
Statistical Analysis 34: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HRW-HPV incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2825). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 5.72, 95% CI 2-sided [5.36 to 6.10]
Statistical Analysis 35: Comparison: Vacc-039 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HR-HPV incident cervical infection, in subjects who participated in the HPV-039 study and who received HPV vaccine in that study (N=2823). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 5.29, 95% CI 2-sided [4.94 to 5.65]
Statistical Analysis 36: Comparison: Vacc-092 Group; Analysis was performed to assess the protective effect of HPV Vaccine in terms of incidence rate of oncogenic HR-HPV incident cervical infection, in subjects who participated in the HPV-039 study and who received placebo in that study (N=2825). Those subjects were or were not enrolled in the current study, were HPV DNA negative subjects at baseline and had cervical samples collected data; Test type: Other — [test comment as in outcome 9, analysis 1]; Incidence rate per 100-Person years = 6.29, 95% CI 2-sided [5.91 to 6.69]

ADVERSE EVENTS:
Time Frame: During the entire study period (Day 1-Month 12)
Description: Other AEs were collected only on the vaccinated subjects in this study (Vacc-092 Group) while SAEs were collected on enrolled subjects of both groups in this study.
Arm/Group | Vacc-039 Group | Vacc-092 Group
All-Cause Mortality (participants affected / at risk) | 0/1671 | 0/1866
Serious Adverse Events (participants affected / at risk) | 0/1671 | 1/1866
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1791
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vacc-039 Group (N=1671) | Vacc-092 Group (N=1866)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vacc-039 Group (N=0) | Vacc-092 Group (N=1791)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT03629886/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03629886/SAP_001.pdf